CLINICAL TRIAL: NCT00480961
Title: Congestive Heart Failure Surgical Treatmment With Autologous Stem Cell Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Mediterranean Institute for Transplantation and Advanced Specialized Therapies (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRRB/00/2006
Record Dates: First submitted 2007-05-31; First posted 2007-06-01 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2007-05

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: intramiocardiac autograft of autologous stem cells

SUMMARY:
This research study was designed to test the safety and effectiveness of autologous stem cell graft in the myocardium of patients with refractory Congestive Heart Failure (CHF) with ischemic etiology. Cellular implantation will take place during off-pump revascularization surgery or during an ad hoc procedure using a mini-thoracotomy access.

DETAILED DESCRIPTION:
Primary target: determine the safety of introducing CD 34+ autologous progenitor cells (centrally grafted or mobilized in peripheral blood) in the myocardium of ischemic cardiac disease patients. Secondary target: determine clinical effects of grafted cells on remodeling pathology.

ELIGIBILITY:
Inclusion criteria

* Age >18 y/o
* CHF with EF > 35%
* Bilirubinemia, serum transaminase> 2.5 times normal max level
* Creatininemia > 2.5 times max level
* NYHA Class > 3
* Negative pregnancy test (for women in fertile age)

Exclusion criteria

* Impossibility to harvest the bone marrow
* Pregnancy or breast-feeding
* History of malignant neoplasia in the 5-year period before the study (save for in-situ carcinoma of the cervix treated successfully and skin tumors - not melanomas)
* Incapability or unwillingness to comply with the envisaged treatment protocol, follow-up, or tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-05

PRIMARY OUTCOMES:
Primary target: determine the safety of introducing CD 34+ autologous progenitor cells (centrally grafted or mobilized in peripheral blood) in the myocardium of ischemic cardiac disease patients. | 1 YEAR

SECONDARY OUTCOMES:
Secondary target: determine clinical effects of grafted cells on remodeling pathology. | 1 YEAR

CONTACTS AND LOCATIONS:
Overall Officials: CESARE SCARDULLA, md, Principal Investigator — The Mediterranean Institute for Transplantation and Advanced Specialized Therapies
Locations (1):
- Ismett, Palermo, pa, Italy